CLINICAL TRIAL: NCT03845855
Title: The Investigation of the Effects of Virtual Reality Training on Dual Task Performance, Balance and Gait on Patients With Chronic Stroke
Brief Title: Effects of Virtual Reality on Dual Task Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Büşra Kayabınar, Lecturer, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018.09.97
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: virtual reality; stroke; dual task
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality with robotic gait (Experimental): virtual reality treatment with robotic gait therapy 2 times for week by 6 weeks.
  Interventions: Other: virtual reality; Other: robotic gait
- Robotic gait therapy only (Active Comparator): only robotic gait therapy 2 times for week by 6 weeks
  Interventions: Other: robotic gait

INTERVENTIONS:
Other: virtual reality — Virtual reality with a game
  Arms: Virtual reality with robotic gait
Other: robotic gait — robotic gait therapy

SUMMARY:
This study evaluates the effects of virtual reality treatment in addition to robotic gait therapy on dual task performance, balance and gait in chronic stroke patients. Half of participants will attend virtual reality treatment in addition to robotic gait therapy for 12 sessions, while the other half will attend only robotic gait therapy for 12 sessions.

DETAILED DESCRIPTION:
Following stroke, motor disorders, balance disorders, falls, gait disturbances and cognitive disorders are frequently seen. In stroke rehabilitation, with the use of robots and virtual reality systems with conventional methods, it is aimed to increase patient's motivation, to check if exercise is effective, to provide objective evaluation data and to support the motor learning process and the use of these methods in the field of neurological rehabilitation is increasing.

Multi-task evaluations can be made with the virtual environments created by virtual reality applications and complex tasks.

The traditional approach to stroke rehabilitation is mainly focused on balance and gait training under single task conditions. In everyday life, people should not only have balance and mobility skills, but also have the ability to perform other cognitive and motor tasks with these skills. Therefore, traditional approaches are not sufficient for the individual to return to society after a stroke.

In this respect, this study was planned in order to examine the effects of frequently used virtual reality treatment in addition to robotic gait therapy on the dual task, balance and gait performance.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research
* Stroke for the first time
* To be able to walk independently before the disease
* To score 3 or above in the functional ambulation classification
* 6 months after stroke diagnosis
* Not having open wounds
* Severity of spasticity of the lower extremities to be 3 and below according to the Modified Asworth Scale
* To score 24 or more in the Mini Mental State Examination

Exclusion Criteria:

* Acute internal problems, additional neurological diseases, or orthopedic problems that might limit walking
* To have received botulinum toxin treatment during 6 months before treatment or during treatment
* To have stroke on both sides
* To have neglect

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
10 meter walk test | change from baseline time at the end of 6 week
  The time is measured after 10 meter walk completed
10 meter walk test with cognitive task | change from baseline time at the end of 6 week
  The time is measured after 10 meter walk with a cognitive task completed
10 meter walk test with motor task | change from baseline time at the end of 6 week
  The time is measured after 10 meter walk with a motor task completed

SECONDARY OUTCOMES:
Mini Mental State Examination | change from baseline score at the end of 6 week
  Mini Mental State Examination can be used to assess the mental status. Mini Mental State Examination is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30. The minimum score is 0. Getting 24 point is cut point. If a person get 24 points from examination, his/her mental status is fine. The higher scores represent better mental status.
Functional Ambulation Classification | change from baseline score at the end of 6 week
  This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. Level 0 is the minimum level and level 5 is the maximum level. Higher levels represent better function.
Rivermead Mobility Index | change from baseline score at the end of 6 week
  Rivermead Mobility Index assesses functional mobility in gait, balance and transfers after stroke. 14-self-reported items and 1 direct observation item are calculated. Items are coded as either 0 or 1, depending on whether the patient can complete the task according to specific instructions. Items receive a score of 0 for a "No" response and 1 for a "Yes" response.A maximum of 15 points is possible; higher scores indicate better mobility performance.
Berg Balance Scale | change from baseline score at the end of 6 week
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Falls Efficacy Scale - International | change from baseline score at the end of 6 week
  The Falls Efficacy Scale International are measures of "fear of falling" or, more properly, "concerns about falling". Minimum 16 (no concern about falling) to maximum 64 (severe concern about falling) can be obtained.
Functional Gait Assessment | change from baseline score at the end of 6 week
  The Funcitonal Gait Assessment is used to assess postural stability during various walking tasks. The highest score is 30/30. Higher scores represent better functional gait performance.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Kayabınar, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Kozakli Fizik Tedavi Ve Rehabilitasyon Hastanesi, Nevşehir, Kozaklı, Turkey (Türkiye)